CLINICAL TRIAL: NCT07306169
Title: Effect of Baduanjin Exercise on the Rehabilitation of Patients With Parkinson's Disease: A Randomized Controlled Study
Brief Title: Baduanjin Qigong Exercise In Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulay karacaoglu, Head of Physiotherapy and Rehabilitation, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/2023-12
Record Dates: First submitted 2025-12-12; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: parkinson; baduanjin; rehabilitation
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial included 27 elderly individuals diagnosed with Parkinson's disease who were living in a nursing home. Participants were randomly assigned to an experimental group (n=13) and a control group (n=14). The experimental group received traditional physiotherapy combined with Baduanjin exercises for three months, while the control group received only traditional physiotherapy. Before and after the intervention, participants were evaluated using the Berg Balance Scale (BBS), Timed Up and Go Test (TUG), Six-Minute Walk Test (6MWT), and the Unified Parkinson's Disease Rating Scale-Motor Examination (UPDRS-III).
Who Masked: Participant
Masking Description: Participant blinding was applied, as individuals did not know which intervention group they belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phsical therapy (Experimental): A modified Parkinson's rehabilitation program suitable for elderly residents was implemented. Sessions were held three times per week for 45 minutes over three months. The program included walking practice, stair climbing, sit-to-stand exercises, backward and toe walking, single-leg stance, tandem and lateral walking, turning, weight-shifting with support, and balance exercises using balls and therabands. Strengthening, gait training to improve step length and directional changes, warm-up walking, and breathing exercises were also incorporated. All sessions were conducted in small groups of 3-4 participants.
  Interventions: Other: physical therapy
- baduanjin exercise (Experimental): A modified Baduanjin program based on the traditional eight movements was applied. The session lasted 15 minutes and each movement was performed for 6-8 repetitions. Exercises included raising the arms in coordination with breathing, a bow-and-arrow movement for scapular control, gentle lateral bending, trunk rotation for postural stability, side leaning for core balance, a forward-reaching movement with bent knees to enhance flexibility, shoulder lifting and releasing for relaxation, and circular arm motions to promote upper-limb mobility and coordination. All movements were adapted to be safe and manageable for older adults.
  Interventions: Other: physical therapy; Other: baduanjin exercise

INTERVENTIONS:
Other: physical therapy — A modified Parkinson's rehabilitation program suitable for elderly residents was implemented. Sessions were held three times per week for 45 minutes over three months. The program included walking practice, stair climbing, sit-to-stand exercises, backward and toe walking, single-leg stance, tandem and lateral walking, turning, weight-shifting with support, and balance exercises using balls and therabands. Strengthening, gait training to improve step length and directional changes, warm-up walking, and breathing exercises were also incorporated. All sessions were conducted in small groups of 3-4 participants.
Other: baduanjin exercise — A modified Baduanjin program based on the traditional eight movements was applied. The session lasted 15 minutes and each movement was performed for 6-8 repetitions. Exercises included raising the arms in coordination with breathing, a bow-and-arrow movement for scapular control, gentle lateral bending, trunk rotation for postural stability, side leaning for core balance, a forward-reaching movement with bent knees to enhance flexibility, shoulder lifting and releasing for relaxation, and circular arm motions to promote upper-limb mobility and coordination. All movements were adapted to be safe and manageable for older adults.
  Arms: baduanjin exercise

SUMMARY:
This study investigates whether adding Baduanjin exercise, a gentle and easy-to-learn traditional Chinese mind-body practice, can contribute to rehabilitation in individuals with Parkinson's disease. Parkinson's disease commonly leads to impairments in balance, walking, and overall motor function, which may affect independence and quality of life.

In this randomized controlled study, participants living in a nursing home were assigned to one of two groups:

a control group receiving standard physiotherapy, and an experimental group receiving Baduanjin exercise in addition to standard physiotherapy for 12 weeks.

Throughout the study, participants were assessed on balance, mobility, walking endurance, and motor symptoms using validated clinical tools.

DETAILED DESCRIPTION:
This randomized controlled study is designed to evaluate the effects of incorporating Baduanjin exercise, a traditional low-intensity mind-body practice, into a standard physiotherapy program for individuals with Parkinson's disease residing in a long-term care facility. Parkinson's disease frequently results in motor impairments such as postural instability, reduced gait speed, decreased walking endurance, and limitations in functional mobility, creating a need for accessible rehabilitative approaches.

Participants who met the inclusion criteria were randomly assigned to one of two groups: (1) a control group receiving conventional physiotherapy alone, or (2) an experimental group receiving Baduanjin exercise in addition to conventional physiotherapy. The intervention lasted 12 weeks. The Baduanjin program consisted of eight simplified movements emphasizing balance, postural control, coordinated breathing, and gentle whole-body mobility. Both groups participated in supervised sessions three times per week.

Outcome measures included standardized clinical assessments of balance, functional mobility, walking endurance, and motor symptom severity. These assessments were conducted at baseline and following completion of the 12-week intervention period to record changes over time.

The purpose of this study is to determine whether integrating Baduanjin into routine physiotherapy is feasible and appropriate as a complementary rehabilitative strategy for individuals with Parkinson's disease living in long-term care settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years and older residing in a nursing home

  * A diagnosis of Parkinson's disease classified as Hoehn & Yahr Stages 1-3
  * Sufficient cognitive ability to follow exercise instructions
  * Willingness to voluntarily participate in the study

Exclusion Criteria:

* Severe dementia or cognitive impairment

  * Unstable cardiovascular disease
  * Significant visual or hearing loss
  * Severe osteoarthritis, recent fractures, or movement limitations
  * Inability to follow instructions in Turkish
  * Inability to continue the exercise program during the study period or withdrawal of informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
balance | through study completion, an average of 6 months
  The Berg Balance Scale is one of the most commonly used tests to assess an individual's balance status. It consists of 14 items, each scored from 0 to 4. Total scores between 0-20 indicate a high risk of falling, 21-40 indicate a moderate fall risk, and 41-56 indicate a low fall risk.
mobility | through study completion, an average of 6 months
  The Timed Up and Go (TUG) Test is used to assess fall risk and mobility in older adults. The test requires a chair and a stopwatch. The patient is asked to stand up from the chair, walk 3 meters, turn, walk back, and sit down again. The time taken to complete the task is recorded as the test result. A completion time greater than 12 seconds indicates an increased risk of falling.
walking capasity | through study completion, an average of 6 months.
  The Six-Minute Walk Test (6MWT) is used to assess functional capacity, which is an important predictor of morbidity and mortality. The distance an individual walks in six minutes is recorded in meters. Reference values include approximately 380 m for individuals with COPD (<160 m indicates increased mortality risk), 590-640 m for adults aged 20-50 years, 540-570 m for those aged 60-70 years, and 470-530 m for individuals aged 70-80 years.
parkinson degree | through study completion, an average of 6 months.
  The Unified Parkinson's Disease Rating Scale (UPDRS), Part III, assesses the motor examination of individuals with Parkinson's disease. During the assessment, the examiner demonstrates each movement while providing instructions and then evaluates the patient's performance. Each item is scored on a scale from 0 to 4, and all motor functions are assessed separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Mudanya University, Bursa, Turkey (Türkiye)